CLINICAL TRIAL: NCT02779595
Title: Change of Regional Ventilation During Spontaneous Breathing After Lung Surgery
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: thoraxEIT
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Infection; Respiratory Insufficiency; Aspiration Pneumonitis; Bronchospasm; Atelectasis
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia, Aspiration; Bronchial Spasm; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung surgery: 26 patients (up to 36) undergoing lung surgery having an elevated risk for postoperative pulmonary complications will be examined by perioperative pulmonary function tests
  Interventions: Other: Perioperative pulmonary function tests
- Flail chest: 8 patients undergoing an operative stabilization of a flail chest will be examined by perioperative pulmonary function tests
  Interventions: Other: Perioperative pulmonary function tests

INTERVENTIONS:
Other: Perioperative pulmonary function tests — Pulmonary electrical impedance tomography, spirometry, pulse oximetry and query performed preoperatively, at the the third, fifth and seventh postoperative day

SUMMARY:
Perioperative changes in regional ventilation by pulmonary electrical impedance tomography and spirometry will be investigated in patients at risk for postoperative pulmonary complications. Those patients undergo lung and flail chest surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (Defined as pulmonary infection, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis or respiratory insufficiency subsequent to surgery) increase the morbidity and mortality of surgical patients. Several independent factors determined by the patients' characteristics and the operative procedure increase the risk for those complications. The postoperative decrease of values measured by spirometry, such as the forced vital capacity (FVC) and forced expiratory volume in one second (FEV1), were found in patients after major surgical procedures for several days. The postoperative reduction of those measurement can be the result of general functional limitations in those patients (e.g. by postoperative pain) or the result of a regional postoperative pulmonary complication (e.g. atelectasis, pleural effusion). The method of the electrical impedance tomography (EIT) enables to visualize the regional ventilation within a transversal section of the lung in real time. Studies examining the change of pulmonary EIT for several days postoperatively in spontaneously breathing patients are lacking. The aim of the present study is to examine perioperative changes in regional ventilation in spontaneously breathing patients during their recovery after lung and flail chest surgery. Moreover, the association of those changes with expected changes in spirometry is tested. Finally, in patients with evident postoperative pulmonary complications the value of pulmonary EIT to detect those changes is investigated. The study should improve the knowledge about the development of postoperative pulmonary complications and test the scientific and clinical value of pulmonary EIT in those spontaneously breathing patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Inpatient
* Lung surgery under general anaesthesia

Exclusion Criteria:

* Missing informed consent
* Outpatient
* Emergency procedure
* Revision surgery of hospitalized patients
* Pneumothorax
* Pleural effusion
* Pleural effusion or pleural empyema with need to cannulate
* scheduled Pneumonectomy
* Expected hospital stay of less than three days
* Pregnancy
* Allergy against material of the electrode belt (silicone rubber, stainless steel, gold-plated brass)
* Injured, inflamed or otherwise affected skin within the target region of the electrode belt
* Unstable spine injury
* Body mass index of more than 50 kg/m2
* Incapacity to lie quietly for the examination
* Pacemaker, defibrillator or other active implant
* Reoperation before the examination at the third postoperative day

Exclusion criteria during clinical course:

* performed pneumonectomy
* Reoperation
* postoperative ventilation at the third day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult inpatients undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Lateral Change from baseline in regional ventilation | baseline and 3. postoperative day
  Regional ventilation is measured by pulmonary electrical impedance tomography. The ipsi- and contralateral change in the calculated 'Center of Ventilation' is evaluated

SECONDARY OUTCOMES:
Lateral Change from baseline in regional ventilation depending on side of surgery | baseline and 3. postoperative day
  Regional ventilation is measured by pulmonary electrical impedance tomography. The influence of the side of surgery on the ipsi- and contralateral change in the calculated 'Center of Ventilation' is evaluated

OTHER OUTCOMES:
Association between lateral change of regional ventilation and change of forced vital capacity | baseline, 3., 5. and 7. postoperative day
  Correlation testing is done on the ipsi- and contralateral change in the calculated 'Center of Ventilation' and the forced vital capacity in % of normal (FVC%) by spirometry
Sagittal change from baseline in regional ventilation | baseline, 3., 5. and 7. postoperative day
  Regional ventilation is measured by pulmonary electrical impedance tomography. The sagittal change in the calculated 'Center of Ventilation' is evaluated
Association between sagittal change of regional ventilation and change of forced vital capacity | baseline, 3., 5. and 7. postoperative day
  Correlation testing is done sagittal change in the calculated 'Center of Ventilation' and the forced vital capacity in % of normal (FVC%) by spirometry
Time shift in regional ventilation between ipsi- and contralateral lung | baseline, 3., 5. and 7. postoperative day
  Regional ventilation is measured by pulmonary electrical impedance tomography. The shift in time of occurence of ipsi- and contralateral Ventilation is evaluated
Impact on flail chest surgery to change from baseline in regional ventilation | baseline, 3., 5. and 7. postoperative day
  Measured by EIT

CONTACTS AND LOCATIONS:
Overall Officials: Markus Kredel, PD.Dr.med, Principal Investigator — University of Würzburg, Department of Anaesthesia and Critical Care
Locations (1):
- University of Würzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Background] Karayiannakis AJ, Makri GG, Mantzioka A, Karousos D, Karatzas G. Postoperative pulmonary function after laparoscopic and open cholecystectomy. Br J Anaesth. 1996 Oct;77(4):448-52. doi: 10.1093/bja/77.4.448. PMID 8942326
- [Background] Guizilini S, Bolzan DW, Faresin SM, Alves FA, Gomes WJ. Ministernotomy in myocardial revascularization preserves postoperative pulmonary function. Arq Bras Cardiol. 2010 Oct;95(5):587-93. doi: 10.1590/s0066-782x2010005000137. Epub 2010 Oct 15. English, Portuguese. PMID 20963310
- [Background] Davoudi M, Farhanchi A, Moradi A, Bakhshaei MH, Safarpour G. The Effect of Low Tidal Volume Ventilation during Cardiopulmonary Bypass on Postoperative Pulmonary Function. J Tehran Heart Cent. 2010 Summer;5(3):128-31. Epub 2010 Aug 31. PMID 23074580
- [Background] Leonhardt S, Lachmann B. Electrical impedance tomography: the holy grail of ventilation and perfusion monitoring? Intensive Care Med. 2012 Dec;38(12):1917-29. doi: 10.1007/s00134-012-2684-z. Epub 2012 Sep 20. PMID 22992946
- [Background] Radke OC, Schneider T, Heller AR, Koch T. Spontaneous breathing during general anesthesia prevents the ventral redistribution of ventilation as detected by electrical impedance tomography: a randomized trial. Anesthesiology. 2012 Jun;116(6):1227-34. doi: 10.1097/ALN.0b013e318256ee08. PMID 22531334
- [Background] Karsten J, Heinze H, Meier T. Impact of PEEP during laparoscopic surgery on early postoperative ventilation distribution visualized by electrical impedance tomography. Minerva Anestesiol. 2014 Feb;80(2):158-66. Epub 2013 Jul 23. PMID 23877309
- [Background] Frerichs I, Hahn G, Golisch W, Kurpitz M, Burchardi H, Hellige G. Monitoring perioperative changes in distribution of pulmonary ventilation by functional electrical impedance tomography. Acta Anaesthesiol Scand. 1998 Jul;42(6):721-6. doi: 10.1111/j.1399-6576.1998.tb05308.x. PMID 9689281
- [Background] Reifferscheid F, Elke G, Pulletz S, Gawelczyk B, Lautenschlager I, Steinfath M, Weiler N, Frerichs I. Regional ventilation distribution determined by electrical impedance tomography: reproducibility and effects of posture and chest plane. Respirology. 2011 Apr;16(3):523-31. doi: 10.1111/j.1440-1843.2011.01929.x. PMID 21261780
- [Background] Guerin C, Frerichs I. Getting a better picture of the correlation between lung function and structure using electrical impedance tomography. Am J Respir Crit Care Med. 2014 Nov 15;190(10):1186-7. doi: 10.1164/rccm.201405-0812IM. No abstract available. PMID 25398109
- [Background] Wrigge H, Zinserling J, Muders T, Varelmann D, Gunther U, von der Groeben C, Magnusson A, Hedenstierna G, Putensen C. Electrical impedance tomography compared with thoracic computed tomography during a slow inflation maneuver in experimental models of lung injury. Crit Care Med. 2008 Mar;36(3):903-9. doi: 10.1097/CCM.0B013E3181652EDD. PMID 18431279